CLINICAL TRIAL: NCT05197244
Title: Randomized Controlled Pilot Study of a Culinary Intervention for Bone Health
Brief Title: A Culinary Intervention for Bone Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB21-1332
Record Dates: First submitted 2021-12-10; First posted 2022-01-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Osteoporosis, Age-Related; Osteoporosis Risk
Keywords: osteoporosis; fracture; culinary nutrition; culinary medicine; teaching kitchen; nutrition
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culinary Medicine Intervention (Experimental): Participants will attend a 2-hour hands-on cooking class in additional to usual care.
  Interventions: Behavioral: Culinary Medicine Intervention
- Control (No Intervention): Participants will receive usual care.

INTERVENTIONS:
Behavioral: Culinary Medicine Intervention — A 2-hour practical culinary medicine program facilitated by a culinary dietitian at a hospital-based teaching kitchen, followed by 3 virtual group follow-up sessions occurring monthly, each lasting approximately 30 minutes. The follow-up sessions will be facilitated by a culinary dietitian and will be conducted using a secure telephone/video conference platform.
  Arms: Culinary Medicine Intervention

SUMMARY:
This is a randomized, controlled pilot study to evaluate the feasibility and acceptability of a single 2-hour culinary medicine intervention for bone health among individuals with age-associated low bone mass.

DETAILED DESCRIPTION:
This is a randomized, controlled pilot study to evaluate the feasibility and acceptability of a single 2-hour culinary medicine intervention for bone health among individuals with age-associated low bone mass. A total of 40 individuals referred to a tertiary osteoporosis centre for age-associated low bone mass will be will be recruited and randomized 1:1 to attend either: 1) a 2-hour hands-on culinary medicine program at a hospital-based teaching kitchen followed by three monthly virtual group meetings, each lasting 30 minutes and led by the facilitator of the culinary nutrition program (intervention group), or, 2) not to attend the culinary nutrition program (control group). Baseline data will be collected at the time of recruitment, and both the intervention and control group will be followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults referred to local tertiary osteoporosis centre for assessment of age-associated low bone mass or assessment of fracture risk
* Women must be postmenopausal (i.e. documented history of surgical menopause, or at least 12 months since last menstrual period), men must be age ≥45 years
* Self-determined ability to learn in classroom and kitchen environments and a virtual (video) learning environment
* Reliable access to hardware, software, and internet connection required to participate in an interactive virtual (video) conference
* Ability to attend local hospital-based teaching kitchen for culinary medicine intervention
* Willing to participate in a culinary medicine intervention and provide informed consent

Exclusion Criteria:

* Complex metabolic bone disease or on dialysis for end-stage kidney disease
* Exclusion on the basis of other active health conditions which may present a contraindication to intake of whole and calcium-rich foods will be determined by the medical team on a case-by-case basis
* Deemed by research team to be unable to learn in a group classroom or kitchen environment
* Unable to communicate in English

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Recruitment capacity | Baseline
  Proportion of total referrals who meet criteria for eligibility screening
Intervention reach | Baseline
  Proportion of eligible individuals who agree to participate in study
Intervention fidelity | 3 months
  Proportion of participants who complete study procedures
Intervention satisfaction | 3 months
  Proportion of the intervention group who indicate that they are satisfied with their experience in the culinary medicine class
Intervention mode and dose | 3 months
  Proportion of the intervention group who would have preferred to attend multiple hands-on culinary medicine sessions rather than a single session

SECONDARY OUTCOMES:
Readiness to change home cooking patterns | Immediately post-intervention
  Proportion of participants who plan to make a change in home cooking patterns
Readiness to change diet | Immediately post-intervention
  Proportion of participants who plan to make a change in diet
Confidence in ability to change home cooking patterns | Immediately post-intervention
  Confidence in ability to change home cooking patterns graded on a scale of 1 (not at all confident) to 10 (very confident)
Confidence in ability to change diet | Immediately post-intervention
  Confidence in ability to change diet graded on a scale of 1 (not at all confident) to 10 (very confident)
Nutrition education needs | Immediately post-intervention
  Proportion of participants requesting additional education regarding nutrition and bone health

OTHER OUTCOMES:
Meals eaten at home | 3 months
  Change in number of meals eaten each week that are prepared at home
Home cooking behaviours | 3 months
  Change in number of meals personally prepared by participant "from scratch" each week
Dietary patterns | 3 months
  Change in weekly intake of fruits, vegetables, dairy (including fermented dairy)
Food skills | 3 months
  Change in score on a modified food skills questionnaire (higher score means better food skills)
Overall diet quality | 3 months
  Change in overall diet quality (assessed using 24-hour food recall)
Dietary calcium intake | 3 months
  Change in daily dietary calcium intake (assessed via 24-hour dietary recall)
Dietary vitamin D intake | 3 months
  Change in daily dietary vitamin D intake (assessed via 24-hour dietary recall)
Dietary protein intake | 3 months
  Change in daily dietary protein intake (assessed via 24-hour dietary recall)
Calcium supplement use | 3 months
  Proportion of participants taking a calcium supplement
Vitamin D supplement use | 3 months
  Proportion of participants taking a vitamin D supplement

CONTACTS AND LOCATIONS:
Overall Officials: Emma O Billington, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No